CLINICAL TRIAL: NCT02739867
Title: Platelet RNA Profiling to Detect Occult Cancer in Patients With Unprovoked Venous Thromboembolism
Brief Title: Tumor-educated Platelets in Venous Thromboembolism
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Harry R. Buller, Professor of Vascular Medicine, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: PLATO-VTE
Record Dates: First submitted 2016-04-12; First posted 2016-04-15 (Estimated); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Neoplasms; Venous Thromboembolism
Keywords: occult cancer; venous thromboembolism; tumor-educated platelets; platelet RNA profiling; early diagnosis; screening
MeSH Terms: conditions — Neoplasms; Venous Thromboembolism; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Platelet pellet, EDTA plasma, citrated plasma, and cell-free DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Unprovoked VTE: Patients aged 40 years or older with a first episode of objectively confirmed, symptomatic, unprovoked deep vein thrombosis of the leg (distal or proximal) or pulmonary embolism

SUMMARY:
Among patients with a first episode of unprovoked venous thromboembolism (VTE), the contemporary one-year risk of detecting occult cancer is approximately 4% to 7%. Of these cases, 30% to 60% are missed by routine limited screening for cancer. RNA profiling of platelets is a promising, highly accurate biomarker for cancer detection, but its clinical utility in patients with unprovoked VTE is unknown. The objective of the present study is to evaluate the diagnostic accuracy of platelet RNA profiling in detecting occult cancer in patients with unprovoked venous thromboembolism. Secondary objectives include evaluation of other biomarkers for cancer, prediction of bleeding, and prediction of recurrent VTE.

ELIGIBILITY:
Inclusion Criteria:

* First episode of objectively confirmed, symptomatic, unprovoked symptomatic pulmonary embolism and/or distal or proximal deep vein thrombosis of the leg
* Age 40 years or older
* Written informed consent

Exclusion Criteria:

* known malignant disease prior to VTE defined as a cancer diagnosis or cancer treatment within the past 5 years (of note: suspected but unconfirmed cancer at diagnosis of VTE is allowed);
* trauma or fracture of the leg, surgical procedures, general anesthesia, or immobilization greater than 3 days within previous 3 months;
* previous unprovoked venous thromboembolism;
* known hereditary or acquired thrombophilia;
* current pregnancy or puerperium (up to 3 months postpartum);
* current estrogen therapy.
* Greater than 10 days after VTE diagnosis;
* Inability for blood withdrawal at baseline;
* Inability or refusal to provide written informed consent.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients of 40 years or older with a first episode of objectively confirmed, symptomatic unprovoked distal or proximal deep vein thrombosis or pulmonary embolism.
Sampling Method: Probability Sample
Enrollment: 476 (Actual)
Dates: Start 2016-06; Primary Completion 2020-10 (Actual); Study Completion 2021-10 (Actual)

PRIMARY OUTCOMES:
Any solid or hematological cancer | Up to one year following venous thromboembolism
  Adjudicated diagnosis of solid or haematological cancer which is confirmed by histology or cytology, or is unequivocally diagnosed by either imaging or tumour markers

SECONDARY OUTCOMES:
Early-stage solid cancer | Up to one year following venous thromboembolism
  Early-stage solid cancer, defined as stage I or II solid cancer according to the American Joint Commissee on Cancer criteria.
Recurrent venous thromboembolism | Up to one year following venous thromboembolism
  Adjudicated recurrent VTE (see full definition in protocol)
Major bleeding | Up to one year following venous thromboembolism
  Adjudicated major bleeding according to the International Society on Thrombosis and Haemostasis criteria
Clinically relevant non-major bleeding | Up to one year following venous thromboembolism
  Adjudicated clinically relevant non-major bleeding according to the International Society on Thrombosis and Haemostasis criteria
Composite of major bleeding and clinically relevant non-major bleeding | Up to one year following venous thromboembolism
All-cause mortality | Up to one year following venous thromboembolism
Cancer-related mortality | Up to one year following venous thromboembolism
Solid cancer | Up to one year following venous thromboembolism
Hematological cancer | Up to one year following venous thromboembolism
Composite of solid cancer and lymphoma | Up to one year following venous thromboembolism

CONTACTS AND LOCATIONS:
Overall Officials: Harry Büller, MD, PhD, Study Chair — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (14):
- KU Leuven, Leuven, Belgium
- Ottawa Hospital, Ottawa, Canada
- Dresden University Clinic, Dresden, Germany
- Italy (4):
  - Bologna University Hospital, Bologna
  - Gabriele D'Annunzio University, Chieti
  - University of Padua, Padua
  - University of Insubria, Varese
- Netherlands (6):
  - Academic Medical Center, Amsterdam, North Holland
  - Flevoziekenhuis, Almere Stad
  - Slotervaartziekenhuis, Amsterdam
  - VU medical center, Amsterdam
  - Tergooiziekenhuizen, Hilversum
  - Leiden University Medical Center, Leiden
- Hospital Universitario Virgen del Rocio, Seville, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Best MG, Sol N, Kooi I, Tannous J, Westerman BA, Rustenburg F, Schellen P, Verschueren H, Post E, Koster J, Ylstra B, Ameziane N, Dorsman J, Smit EF, Verheul HM, Noske DP, Reijneveld JC, Nilsson RJA, Tannous BA, Wesseling P, Wurdinger T. RNA-Seq of Tumor-Educated Platelets Enables Blood-Based Pan-Cancer, Multiclass, and Molecular Pathway Cancer Diagnostics. Cancer Cell. 2015 Nov 9;28(5):666-676. doi: 10.1016/j.ccell.2015.09.018. Epub 2015 Oct 29. PMID 26525104